CLINICAL TRIAL: NCT01787344
Title: Double-blinded, Randomized, Active Control Comparative, Multicenter-designed, Phase III Clinical Trial to Evaluate the Safety and Efficacy of "Botulax®" Versus "Botox®" in Children With Cerebral Palsy
Brief Title: Phase III Clinical Trial of "Botulax®" to Treat Children With Cerebral Palsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hugel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HG-11-02
Record Dates: First submitted 2013-02-05; First posted 2013-02-08 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Other Infantile Cerebral Palsy
Keywords: Other Infantile Cerebral Palsy
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Botulinum toxin type A (Botulax®) (Experimental): Botulinum toxin type A (Botulax®)
  Interventions: Drug: Botulinum toxin type A(Botulax®)
- Botulinum toxin type A(Botox®) (Active Comparator): Botulinum toxin type A(Botox®)
  Interventions: Drug: Botulinum Toxin Type A(Botox®)

INTERVENTIONS:
Drug: Botulinum Toxin Type A(Botox®) — Single administration, 4units/kg body weight dose in patients with hemiplegia, 6units/kg body weight dose in patients with diplegia, Maximum dosage 200units
  Arms: Botulinum toxin type A(Botox®)
Drug: Botulinum toxin type A(Botulax®) — Single administration, 4units/kg body weight dose in patients with hemiplegia,6units/kg body weight dose in patients with diplegia, Maximum dosage 200units
  Arms: Botulinum toxin type A (Botulax®)

SUMMARY:
To compare the safety and efficacy of Botulax Inj.®(Botulinum toxin type A, Hugel, South Korea) with Botox Inj.® (Botulinum toxin type A, Allergan, USA) in the treatment of cerebral palsy in children.

ELIGIBILITY:
Inclusion Criteria:

1. Children patients ages from 2years old to 10years old.
2. Patients who diagnosed with cerebral palsy.
3. Patients who diagnosed as Gross Motor Function Classification System level I, II, or III
4. Patients who diagnosed as dynamic equinus foot deformity
5. Patients who agree with participation and signed to written agreement by substitute. (Get a signature from children patients if possible)deformity and I, II or III level of Gross Motor Function Classification System

Exclusion Criteria:

1. Patients who had previous injection of other botulinum toxin products in 3 months
2. Patients with hypersensitivity history to botulinum toxin products previously
3. Patients with neuromuscular junction disorder (myasthenia gravis, Lambert- Eaton syndrome, or amyotrophic lateral sclerosis, etc.)
4. Those who have severe cardiovascular, kidney, liver, or respiratory diseases
5. Those who are taking anticoagulant drugs or have bleeding disorder.
6. Pratients with treatment of following drugs: Anticonvulsants, tranquilizers, narcotics, aminoglycoside antibiotics, muscle relaxtants like baclofen, blockers of parasympathetic nervous system, and levodopa.
7. Patients who had history of surgery, plan to have surgery on legs, foot, or ankle.
8. Patients who have evidence of fixed contractures regarding to Investigator
9. Patients who have difference between two legs over 5cm
10. Patients with severe athetoid movement
11. Patients who had other treatments related to dynamic equinus foot deformity, such as alcohol injection or muscle relaxants
12. Those who were not enrolled in other studies within 30 days, or were not paseed over 5 times of half life for clinical trial drugs.
13. Patients who have possibility to take prevented drugs
14. Subjects who are not eligible for this study based on investigator's judgement

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 144 (Actual)
Dates: Start 2012-03; Primary Completion 2014-06 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Rate of patients with an improvement more than two grade in Physician's Rating Scale score. | at 12 weeks post-injection

SECONDARY OUTCOMES:
Rate of patients with an improvement more than two grade in Physician's Rating Scale score, comparing to baseline. | at 6 and 24weeks post-injection
Rate of change in Passive range of motion, compare to baseline. | at 6, 12 and 24 weeks post-injection
Rate of change in Gross Motor Function Measure 88, 66, compare to baseline. | at 6, 12 and 24 weeks post-injection
Rate of change in Modified Tardieu Scale(Ankle DF), compare to baseline. | at 6, 12 and 24 weeks post-injection

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-yi Kwon, M.D., Ph.D., Study Chair — Samsung Medical Center -Seoul
Locations (6):
- South Korea (6):
  - St. Vincent's hospital, Suwon, Kyunggi
  - Samsung medical center - Changwon, Changwon
  - Keimyung University Dongsan Medical Center, Daegu
  - Catholic university of Korea, Daejeon St. Mary's hospital, Daejeon
  - Samsung medical center - Seoul, Seoul
  - The Catholic University of Korea, Seoul St. Mary's hospital, Seoul